CLINICAL TRIAL: NCT03629743
Title: Correlate of Surface Electroencephalogram (EEG) With Implanted EEG Recordings (ECOG)
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David R. Drover, Principle Investigator, Stanford University
Other Study IDs: 45987
Record Dates: First submitted 2018-05-29; First posted 2018-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ECOG and EEG Sensor: Study subjects are neurosurgical patients with medically refractory epilepsy who will have implanted with intracranial ECoG electrodes. The electrodes will be used during a period of inpatient monitoring to identify resectable seizure foci.
  Interventions: Device: EEG; Device: ECOG

INTERVENTIONS:
Device: EEG — EEG will be collected with Brain Product's VAMP-16 channel EEG Monitor using the accompanying software. (Website with further specifications and product details: https://www.brainproducts.com/productdetails.php?id=15)
Device: ECOG — ECOG will be collected with Nihon Kohden acquisition System and accompanying software and depth electrodes.

SUMMARY:
Improve understanding of the correlation between surface EEG and implanted EEG recordings

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects 18 years of age or older.
* English or Spanish Speaking
* Subjects who have been previously diagnosed with intractable epilepsy and require implantation of invasive electrophysiological recordings as part of their routine clinical presurgical workup.

Exclusion Criteria:

* Patients with skin abnormalities at the planned application sites that would interfere with sensor or electrode applications.
* Patients with pre-existing conditions and/or co-morbidities that would prohibit them from participating in the study due to unacceptable risks to their health and well-being, as determined by the Principal Investigator (PI).
* Patients who the PI deems ineligible at the PI's discretion
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stanford Health Care and Clinics
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram (EEG) change before, during, and after anesthesia. | Up to 48 hours. Specific time points are dependent on patient clinical events.
  Patient subjective level of consciousness during and after anesthesia administration will be assessed using response to verbal stimuli, response via button press, reported subjective level of consciousness, and/or response to memory tests (i.e. demonstration of explicit memory recall). Around loss and recovery of consciousness time points (e.g. induction or emergence from anesthesia or when patient falls asleep or wakes up during 24 hour postoperative time points) level of consciousness will be assessed in brief intervals (seconds) until patient no longer responds or begins to respond. Data collected before, after, and during seizure activity if a patient loses consciousness or has diminished consciousness may also be compared.

SECONDARY OUTCOMES:
Electrocardiogram (EEG) change during any changes in consciousness. | Up to 48 hours. Specific time points are dependent on patient clinical events.
  Scalp and cortical electrical activity collected using EEG and ECOG arrays respectively will be analyzed using standard frequency-derived measures (e.g. spectrograms, Fourier analysis), nonlinear dynamical analyses (e.g. correlation dimension, entropy), network dynamics (e.g. connectivity matrices, path length), and/or machine learning. These measures will include all of the data collected from the start of the implant procedure until 24 hours after the implant procedure has ended. Data collected before, after, and during seizure activity if a patient loses consciousness or has diminished consciousness may also be compared. Reports will included characterization of electrophysiological activity before, during, and after variations in behavioral and subjectively reported consciousness.
Electrocardiogram (EEG) change during any seizures. | Up to 48 hours. Specific time points are dependent on patient clinical events.
  Scalp and cortical electrical activity collected using EEG and ECOG arrays respectively will be analyzed using standard frequency-derived measures (e.g. spectrograms, Fourier analysis), nonlinear dynamical analyses (e.g. correlation dimension, entropy), network dynamics (e.g. connectivity matrices, path length), and/or machine learning. Data collected before, after, and during seizure activity if a patient loses consciousness or has diminished consciousness may also be compared. Reports will include characterization and comparison of EEG and ECOG electrophysiological activity and analyses during consciousness transitions and significant time points.

CONTACTS AND LOCATIONS:
Overall Officials: David Drover, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hashiguchi K, Morioka T, Yoshida F, Miyagi Y, Nagata S, Sakata A, Sasaki T. Correlation between scalp-recorded electroencephalographic and electrocorticographic activities during ictal period. Seizure. 2007 Apr;16(3):238-47. doi: 10.1016/j.seizure.2006.12.010. Epub 2007 Jan 19. PMID 17236792
- [Background] Asano E, Brown EC, Juhasz C. How to establish causality in epilepsy surgery. Brain Dev. 2013 Sep;35(8):706-20. doi: 10.1016/j.braindev.2013.04.004. Epub 2013 May 15. PMID 23684007
- [Background] Smith EH, Liou JY, Davis TS, Merricks EM, Kellis SS, Weiss SA, Greger B, House PA, McKhann GM 2nd, Goodman RR, Emerson RG, Bateman LM, Trevelyan AJ, Schevon CA. The ictal wavefront is the spatiotemporal source of discharges during spontaneous human seizures. Nat Commun. 2016 Mar 29;7:11098. doi: 10.1038/ncomms11098. PMID 27020798
- [Background] Ramantani G, Maillard L, Koessler L. Correlation of invasive EEG and scalp EEG. Seizure. 2016 Oct;41:196-200. doi: 10.1016/j.seizure.2016.05.018. Epub 2016 Jun 10. PMID 27324839
- [Background] Hajat Z, Ahmad N, Andrzejowski J. The role and limitations of EEG-based depth of anaesthesia monitoring in theatres and intensive care. Anaesthesia. 2017 Jan;72 Suppl 1:38-47. doi: 10.1111/anae.13739. PMID 28044337
- [Background] Fahy BG, Chau DF. The Technology of Processed Electroencephalogram Monitoring Devices for Assessment of Depth of Anesthesia. Anesth Analg. 2018 Jan;126(1):111-117. doi: 10.1213/ANE.0000000000002331. PMID 28786839
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092